

## Health Economics Research Centre

## Nuffield Department of Population Health

Old Road Campus, Roosevelt Drive, Headington, Oxford OX3 7LF, UK

Tel: +44 (0)1865 289272/3

E-mail: herc@dph.ox.ac.uk

| | Study Code: | ly Code: Participant identification number: | | er: | | | | |
|---|---|---|---|---|---|---|---|---|
| | CONSENT FORM | | | | | | | |
| | Study: Type-2 diabetes: risk perceptions and self-management behaviour | | | | | | | |
| | Researcher: Thomas Rouyard | | | | | | | |
| | | | | | | If you | agree, plea | ase initial box |
| 1. | I confirm that I have read the information sheet dated 29 March 2017 (version 3) for this study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | | | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | | | | | |
| 3. | . I understand that data collected during the study may be looked at by individuals from University of Oxford, from regulatory authorities [and from the NHS Trust(s)], where it is relevant to my taking part in this research. I give permission for these individuals to have access to these data. | | | | | | | |
| 4. | I agree to my General | Practitioner being in | forme | d of my p | articipatio | on in the s | study. | |
| 5. | I understand that the form to support other re | | | - | | | • | |

| Name of Participant | Date | Signature | Signature |
|-------------------------------|------|-----------|-----------|
| Name of Person taking Consent | | Signature | |

Consent Form \_ version 1.0

Type-2 diabetes: risk perceptions and self-management behaviour

Thomas Rouyard

by it.

6. I agree to take part in this study.

IRAS project ID: 210623 1

7 April 2017

<sup>\*1</sup> copy for participant; 1 copy for researcher site file; 1 (original) to be kept in medical notes (if participant is a patient).